CLINICAL TRIAL: NCT07018245
Title: A Phase II, Randomized, Double-Blind, Multi-Center, Placebo-Controlled, Parallel-GroupClinical Trial to Evaluate the Safety and Efficacy of TJ0113 Capsules in Patients withDepressive Disorder
Brief Title: Clinical Trial of TJ0113 Capsules in the Treatment of Patients With Depressive Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou PhecdaMed Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJJS01-101
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TJ0113 200mg (Experimental): Subjects will receive 200 mg of TJ0113 capsules for 8 consecutive weeks
  Interventions: Drug: TJ0113
- TJ0113 400mg (Experimental): Subjects will receive 400 mg of TJ0113 capsules for 8 consecutive weeks
  Interventions: Drug: TJ0113
- Placebo (Placebo Comparator): Subjects will receive 200mg or 400 mg of placebo for 8 consecutive weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TJ0113 — 200 mg or 400 mg Capsule, Once Daily
  Arms: TJ0113 200mg; TJ0113 400mg
Drug: Placebo — Capsule, Once Daily
  Arms: Placebo

SUMMARY:
This study is a phase II, randomized, double-blind, multi-center, placebo-controlled, parallel-group clinical trial and 150 subjects with depressive disorder will be enrolled. Subjects will be randomly assigned in a 1:1 ratio to two cohorts (Cohort 1: 200 mg dose group; Cohort 2: 400 mg dose group). Within each cohort, subjects will be randomized in a 2:1 ratio to either the TJ0113 capsule group or the placebo group, with approximately 50 subjects receiving TJ0113 capsules and approximately 25 receiving placebo. Approximately 50 subjects will be enrolled in each of the TJ0113 capsule 200 mg group, TJ0113 capsule 400 mg group, and placebo group in this trial. Eligible subjects will be randomly assigned to receive continuous oral administration for 8 weeks, after which efficacy and safety will be evaluated, followed by an additional 1-week follow-up period after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily participates in the trial and signs the informed consent form (ICF);
2. Male or female subjects, aged between 18 and 65 years (inclusive) at the time of signing ICF;
3. Subjects whose HAMD-17 score ≥18 during the screening and baseline periods;
4. Subjects who meet the diagnostic criteria for depressive disorder as defined in the Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition) (DSM-5), without psychotic symptoms;
5. Subjects whose Clinical Global Impressions-Severity (CGI-S) scores ≥4 during the screening and baseline periods;
6. Subjects who agree to discontinue the use of other antidepressants, anxiolytics, antipsychotics, mood stabilizers, benzodiazepine sedative-hypnotics, etc., except those specified in the study protocol during the treatment period; Subjects with reproductive potential (including spouses of male subjects) must have no plans for pregnancy or sperm donation from the screening period until 6 months after the last dose and must be willing to use at least one effective contraceptive method (such as abstinence, condoms, etc., as detailed in Section 5.3).

Exclusion Criteria:

1. Presence of any medical condition that may interfere with the participation in the trial, including but not limited to the following: history of malignant tumors, history of epilepsy or complications, hemolytic anemia, pulmonary embolism, or respiratory depression;
2. Within 6 months prior to screening, occurrence of congestive heart failure classified as New York Heart Association (NYHA) Class III or higher, unstable angina, acute myocardial infarction, hemorrhagic stroke (stroke), or ischemic stroke (including transient ischemic attack); or undergoing percutaneous coronary intervention, coronary artery bypass grafting, cardiac valve repair/replacement; or presence of severe arrhythmia as determined by the investigator at screening;
3. A personal or family history of long QT syndrome, a family history of sudden death in first-degree relatives (parents, offspring, and siblings) before the age of 40; and/or a personal history of unexplained syncope within 1 year prior to screening; and/or QTcF >450 ms (male) or QTcF >470 ms (female) based on resting ECG results at screening;
4. Patients with uncontrolled hypertension at screening, defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg (checked prior to randomization);
5. Subjects with clinically significant hepatic impairment, defined as total bilirubin (TBIL) >2× the upper limit of normal (ULN) or alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2×ULN;
6. Subjects with clinically significant renal impairment (creatinine clearance [Ccr] <30 mL/min). The Ccr calculation formula is provided in Note b.
7. Subjects with history of any psychiatric disorders other than DSM-5 depressive disorder, including but not limited to: bipolar and related disorders, obsessive-compulsive and related disorders, trauma- and stressor-related disorders, schizophrenia, anxiety disorders, sleep-wake disorders, substance-related and addictive disorders, or depressive episodes secondary to other psychiatric or somatic conditions;
8. Subjects whose HAMD-17 score at baseline shows a reduction ≥25% compared to the screening period.
9. Subjects at risk of suicide: Those who have exhibited suicidal behavior (including actual attempts, interrupted attempts, or failed attempts) within 1 year prior to the first dose, or subjects with a score ≥3 on item 3 (SUICIDE) of the HAMD-17 scale at screening or baseline, or a 'yes' response to items 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) for suicidal ideation, or subjects with a history of suicidal intent/self mutilation behavior during the current depressive episode;
10. Subjects with history or current episode of failure to respond to two adequate courses of antidepressant treatment;
11. Subjects who are receiving systemic psychotherapy (interpersonal therapy, psychodynamic therapy, cognitive behavioral therapy, etc.), music therapy, exercise therapy, acupuncture, or other treatments during screening and/or at baseline, and who will continue to require these treatments during this study period;
12. Subjects who have received electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), vagus nerve stimulation (VNS), deep brain stimulation (DBS), light therapy, etc., within 3 months prior to screening, or are considered by the investigator to currently require such treatment;
13. Subjects who discontinued psychotropic medications less than 5 half-lives before randomization (at least 2 weeks for monoamine oxidase inhibitors and at least 4 weeks for fluoxetine);
14. Subjects with history of severe allergies, or known hypersensitivity/allergic reaction or intolerance to any component of the investigational drug;
15. Subjects with evidence of alcohol abuse (average weekly consumption ≥14 units of alcohol, where 1 unit ≈ 360 mL of beer, 45 mL of spirits, or 150 mL of wine) or alcohol dependence within the 6 months prior to screening, which the investigator considers may interfere with the subject's understanding or completion of the trial;
16. Subjects with history of drug dependence/drug abuse within the past 1 year;
17. Subjects with history of hepatitis B, or positive hepatitis B virus surface antigen (HBsAg) at screening, or positive hepatitis C virus (HCV) antibody, or positive Human immunodeficiency virus (HIV) antibody, or positive treponema pallidum antibody;
18. Subjects who participated in a clinical trial involving the administration of investigational drugs (new chemical entities), devices, or surgical procedures within 3 months or 5 half-lives (whichever is longer) prior to screening;
19. Females with positive pregnancy test during screening or baseline visits, females who are pregnant, breastfeeding, or planning to become pregnant during the trial, or males or females of childbearing potential unwilling to use effective contraception within 6 months after the last dose;
20. Subjects who are unable to swallow medications, or as judged by the investigator, have any condition that may significantly affect drug absorption, distribution, metabolism, and excretion (such as active intestinal disease, partial or complete intestinal obstruction, chronic diarrhea, etc.), or any condition that may pose a hazard to the participating subjects;
21. Subjects with history of organ transplantation (excluding corneal transplantation);
22. Subjects who donated blood or experienced blood loss ≥400 mL, or received blood transfusion within 3 months prior to screening;
23. Subjects with poor compliance or other reasons that make the subject unsuitable for participation in this trial, as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Rating Scale-17 Item Version (HAMD-17) score at 8 weeks post-treatment | After 8 weeks of treatment
  The total score of the HAMD-17 ranges from 0 to 52, with higher scores indicating a more severe degree of depressive symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Shaohua Hu, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No